CLINICAL TRIAL: NCT01821508
Title: Prospective, Open,Randomized, Unicentre Study Comparing Roux-en-Y Gastric Bypass With the Best Clinical Treatment Regarding Improvement of Microvascular Complications of Type 2 Diabetes Mellitus in Obese Patients.
Brief Title: Clinical Study on Metabolic Surgery Compared to the Best Clinical Treatment in Patients With Type 2 Diabetes Mellitus
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Alemão Oswaldo Cruz (Other)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Principal Investigator, Ricardo Vitor Cohen, MD, MD, PhD, Hospital Alemão Oswaldo Cruz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOMS
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Complications of Diabetes Mellitus
Keywords: Gastroplasty, Diabetes Mellitus Type II, Obesity
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus, Type 2; Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical treatment (Active Comparator): Best and most modern clinical treatment of type 2 diabetes mellitus.
  Interventions: Other: Clinical Treatment
- Roux-En-Y gastric bypass surgery (Active Comparator): A "metabolic" surgery consists of any surgical procedure in which there is any anatomical alteration in the gastrointestinal tract by means of a diversion of food passage, resulting in improved metabolic control in patients with type 2 diabetes mellitus [SCHULMAN, 2009].
  Interventions: Procedure: Roux-En-Y gastric bypass surgery

INTERVENTIONS:
Other: Clinical Treatment — metabolic surgery for diabetes and weight control
  Other Names: lifestyle changes for obesity
  Arms: Clinical treatment
Procedure: Roux-En-Y gastric bypass surgery — laparoscopic surgical procedure with Endoscopic Surgical Stapler
  Arms: Roux-En-Y gastric bypass surgery

SUMMARY:
This is a prospective, open, randomized study involving 100 patients with microvascular complications of type 2 diabetes mellitus and obesity, who will undergo gastric bypass (Roux-en-Y gastric bypass ARM A) or receive best medical treatment (ARM B, control arm).

The aim of this study is to evaluate the effects of Roux-en-Y gastric bypass in the control of diabetic nephropathy in diabetic patients with BMI between 30 and 35 kg/m2.

The medical community is confronted with many different studies using various methodologies to investigate the best pharmacological treatment for type 2 diabetes mellitus. The treatment algorithm offers several different options according to the stage of the disease (which is different in each study). In addition, new drugs are being developed over the years, but are not always a guarantee of effective type 2 diabetes mellitus control [MENDES, 2010]. Furthermore, these drugs do not prevent the development of this disease, consequently increasing the risks of microvascular and macrovascular complications.

Conversely, there is considerable evidence that surgery can be an adequate tool to promote type 2 diabetes mellitus remission in patients who are unresponsive to clinical treatment. Gastric bypass surgery is one of the most popular bariatric surgeries in the world, but its effects on microvascular and macrovascular complications of type 2 diabetes mellitus have not been established. Specialists suggest that the rapid and uncontrollable decrease in blood glucose adds to the concern that the surgery may paradoxically cause exacerbation of microvascular complications [LEOW, 2005], whereas gradual improvement in blood glucose before gastric bypass surgery may prevent this paradoxical worsening, leading to an interruption of this process, or even retinopathy, nephropathy, and neuropathy remission.

However, there are no studies comparing the results of these two types of treatment (clinical vs. surgical) in a similar population and assessing the development of microvascular complications of type 2 diabetes mellitus. Therefore, in order to clarify such doubts, it is necessary and extremely desirable to conduct a randomized controlled trial comparing gastric bypass with the best and most modern clinical treatment. Its findings could have a direct impact on hundreds of millions of diabetics by allowing the inclusion of surgical treatment as a safe and feasible therapeutic option for a significant portion of these patients.

DETAILED DESCRIPTION:
Intervention of Roux-En-Y gastric bypass surgery versus best medical treatment in control or reduces microvascular complications such as retinopathy, microalbuminuria and neuropathic.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adult patients with microalbuminuria (more than 30 mg and less than 300 mg or more of urinary albumin per 24 hours), with or without other microvascular complications of type 2 diabetes mellitus, receiving pharmacological treatment for the disease, which may or may not include the use of insulin.
* Age between 18-65 years
* BMI between 30 and 35 Kg/m2
* 15-year or less after type 2 diabetes mellitus diagnosis
* Negative anti-glutamic acid decarboxylase
* Fasting C-peptide higher than 1 ng/ml, increasing in the postprandial period (two hours after mixed meal, ENSURE plus approximately 500 Kcal)

Exclusion Criteria:

* Patient's refusal to participate
* Autoimmune diabetes mellitus
* Previous abdominal surgeries that may make surgery more difficult, increasing the surgical risk
* Previous malabsorptive and restrictive surgeries
* Pregnant women and nursing mothers
* Recent history of neoplasia (< 5 years), except for non-melanoma skin neoplasms
* History of liver disease - liver cirrhosis -, active chronic hepatitis, active hepatitis B and hepatitis C
* Malabsorptive syndromes and inflammatory bowel disease
* Cardiovascular event (acute myocardial infarction, acute coronary syndrome, angioplasty, or bypass in the last 6 months)
* Angina
* Pulmonary embolism or severe thrombophlebitis in the last 2 years
* Positive HIV serum testing
* Psychiatric disorders, including dementia, active psychosis, severe depression, history of suicide attempts, use of illicit drugs, and excessive alcohol consumption in the last 12 months
* Uncontrolled coagulopathy
* Patients with severe retinopathy, nephropathy, and neuropathy (defined as high risk/advanced proliferative retinopathy or amaurosis; stage 5 of chronic kidney disease defined by glomerular filtration rate, patients who need dialysis or renal transplantation; stage 3 of peripheral neuropathy)
* Patients who participated in other clinical trials in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04-18 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the proportion of patients that present normalization of the albumin/creatinine ratio in isolated urine samples (normal value considered as an albumin/creatinine ratio of less than 30 μg/mg ). | 12, 24 and 60 months
  Number of participants achieving remission Titrating the relation of urinary albumin/creatinine

SECONDARY OUTCOMES:
Changes in diabetic retinopathy | 12, 24 and 60 months
  Number of patients achieving resolution or reduction in the degree of retinopathy and/or macular oedema (severity scale)
Changes in diabetic peripheral neuropathy | 12, 24 and 60 months
  Number of patients with new or worsening of neuropathy
Use of pharmacological therapy for type 2 diabetes mellitus | 12, 24 and 60 months
  Number of medications necessary for targeting euglycaemia
Glycemic control | 12, 24 and 60 months
  Number of patients achieving fasting glucose level < 100 and HbA1c < 6.5%
Blood pressure control | 12, 24 and 60 months
  Number of patients achieving systolic blood pressure <130 mm Hg and diastolic <80 mm Hg
Lipids control | 12, 24 and 60 months
  Number of patients with LDL<100 or <70 mg/dL in patients with previous cardiovascular events; HDL>50 mg/dL and triglycerides <150 mg/dL
Quality of life (SF-36) | 12, 24 and 60 months
  SF-36 questionnaire
Changes in hepatic fibrosis | 12, 24 and 60 months
  Reduction of hepatic elastographic resistance

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo V Cohen, MD. PhD, Principal Investigator — Hospital Alemão Oswaldo Cruz
Locations (1):
- Hospital Alemão Oswaldo Cruz, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cohen RV, Pereira TV, Aboud CM, Zanata Petry TB, Lopes Correa JL, Schiavon CA, Pompilio CE, Quirino Pechy FN, Calmon da Costa Silva AC, Cunha da Silveira LP, Paulo de Paris Caravatto P, Halpern H, de Lima Jacy Monteiro F, da Costa Martins B, Kuga R, Sarian Palumbo TM, Friedman AN, le Roux CW. Gastric bypass versus best medical treatment for diabetic kidney disease: 5 years follow up of a single-centre open label randomised controlled trial. EClinicalMedicine. 2022 Nov 11;53:101725. doi: 10.1016/j.eclinm.2022.101725. eCollection 2022 Nov. PMID 36467457
- [Derived] Cohen RV, Pereira TV, Aboud CM, Petry TBZ, Lopes Correa JL, Schiavon CA, Pompilio CE, Pechy FNQ, da Costa Silva ACC, de Melo FLG, Cunha da Silveira LP, de Paris Caravatto PP, Halpern H, Monteiro FLJ, da Costa Martins B, Kuga R, Palumbo TMS, Docherty NG, le Roux CW. Effect of Gastric Bypass vs Best Medical Treatment on Early-Stage Chronic Kidney Disease in Patients With Type 2 Diabetes and Obesity: A Randomized Clinical Trial. JAMA Surg. 2020 Aug 1;155(8):e200420. doi: 10.1001/jamasurg.2020.0420. Epub 2020 Aug 19. PMID 32492126
- [Derived] Cohen RV, Pereira TV, Aboud CM, Caravatto PP, Petry TB, Correa JL, Schiavon CA, Correa M, Pompilio CE, Pechy FN, le Roux CW; MOMS Study Investigators. Microvascular Outcomes after Metabolic Surgery (MOMS) in patients with type 2 diabetes mellitus and class I obesity: rationale and design for a randomised controlled trial. BMJ Open. 2017 Jan 11;7(1):e013574. doi: 10.1136/bmjopen-2016-013574. PMID 28077412